CLINICAL TRIAL: NCT06429475
Title: Anti-Inflammatory Reliever Therapy for Asthma Using Inhaled Budesonide/Formoterol As-needed With or Without Maintenance in South African Children: A Pragmatic Open Label Phase 3 Randomised Controlled Trial
Brief Title: Anti-Inflammatory Reliever South Africa
Acronym: AIRSA001
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREC/00005663/2023
Record Dates: First submitted 2024-04-08; First posted 2024-05-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: asthma; budesonide/formoterol; beclomethasone; budesonide; children; adolescents
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Standard of Care; Beclomethasone; Budesonide; Albuterol

STUDY DESIGN:
Intervention Model Description: Randomised Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- budesonide/formoterol group (Experimental): Budesonide-formoterol fumarate dihydrate at two dose strengths 80/4.5 and 160/4.5 administered via a pressurized metered dose inhaler (pMDI) or dry powder inhaler (DPI), respectively. The dosing will be dependent on asthma symptom severity ranging from 1 dose as needed and titrated up or down depending on asthma control.
  Interventions: Drug: Budesonide/formoterol
- comparator: standard of care group (Active Comparator): Standard of care
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: Budesonide/formoterol — The Investigational Medicinal Product (IMP) consists of a combination of Budesonide (corticosteroid) and Formoterol Furamate (fast-acting β2 agonist) dihydrate. The IMP is currently available and registered in dry powder form turbuhaler (Symbicort) and a pressurised metered dose inhaler (Vannair).
  The recommended doses are pMDI/DPI 80/4.5 1-2 puffs twice daily OR 1 puff as needed (a maximum daily dose of 8 puffs) for children 6-11 years of age and 160/4.5 1-2 inhalations twice daily or 1 puff as needed (a maximum daily dose of 12 puffs) for adolescents 12-18 years.
  Other Names: No other intervention names
  Arms: budesonide/formoterol group
Drug: standard of care — Any therapy that is prescribed as per asthma guidelines i.e. beclomethasone, budesonide and salbutamol, montelukast etc
  Other Names: beclomethasone or budesonide & salbutamol or mentelukast
  Arms: comparator: standard of care group

SUMMARY:
This is a Phase 3 single-centre open label randomised controlled trial with two equal sized groups to assess the efficacy of budesonide/formoterol 80/4.5 (6-11 years) and 160/4.5 (12-18 years) compared to the standard of care in reducing asthma exacerbations over 52 weeks.

Children and adolescents with a diagnosis of asthma or newly diagnosed with asthma will be screened for eligibility for enrolment. Those who had an asthma exacerbation in the previous year will be randomised 1:1, to either receive budesonide/formoterol inhaler for both symptom relief and for chronic anti- inflammatory maintenance therapy or the standard of care which is separate inhalers for symptom relief (short acting bronchodilator salbutamol) and chronic maintenance therapy with inhaled corticosteroids (beclomethasone or budesonide) and/or long-acting beta agonists or montelukast as determined by treating physicians. All asthma exacerbations and clinic/hospital admissions will be recorded for the duration of the 52-week follow-up. Participants will be followed up at 13, 26, 39 and 52 weeks. The 13- and 39-week visit will be telephonic visits to capture the primary end-point i.e. asthma exacerbations. Adverse events and medication changes data will also be collected.

An independent Data and Safety Monitoring Board (DSMB) will be convened for this study with expertise in asthma and asthma clinical trials. The purpose of the DSMB will be to monitor the study for safety and operational futility with pre-defined stopping criteria. In addition, a Trial Steering Committee (TSC) will also provide overall supervision of the trial and ensure the trial is delivered in accordance with ICH-GCP. The TSC has been established with an independent Chair and include additional independent members including an observer early career researcher. Representatives of the Trial Funder (NIHR) and Sponsor (AHRI) will be invited to all TSC meetings.

DETAILED DESCRIPTION:
Over the last two decades non-communicable diseases (NCDs) have been rising in sub-Saharan Africa, and NCDs are set to overtake communicable, maternal, neonatal, and nutritional diseases combined as the leading cause of mortality in sub-Saharan Africa by 2030. Many NCDs have their roots in childhood with lifestyle changes in combination with an increasing median population age in Africa making a further dramatic rise in NCDs in Africa's near future highly likely. The World Health Organization (WHO) now considers the prevention and control of NCDs as an urgent development issue and essential to the achievement of the Sustainable Development Goals (SDG) and this can only be achieved with childhood interventions. The 2018 WHO report on NCDs, reported 3.8 million deaths annually from non-communicable respiratory diseases (asthma and chronic obstructive pulmonary disease), with 78% of deaths in low-income and middle-income countries (LMICs). Asthma morbidity and mortality are preventable with inhaled therapies-however, there is lack of evidence on how to deliver these in an affordable and effective way.

The WHO highlights asthma as an under-appreciated cause of poverty in LMICs that retards economic and social development, erodes the health and well-being of those affected and has a negative impact on families and societies. Asthma aggravates poverty and poverty aggravates asthma. Children miss out on education, adults lose days at work and the costs of drugs, emergency visits, and hospitalization are major financial burdens, not only for individuals/families but also for struggling health systems.

In South Africa, asthma is the most common NCD in childhood affecting 1 in 5 children with a prevalence of asthma symptoms at 21% in adolescence. Despite the availability of asthma medicines in the Essential Medicines List, asthmatic children report having severe asthma symptoms in over 50% of those with asthma. South Africa still reports the fourth highest mortality rate globally. The core to asthma management includes use of chronic use of anti-inflammatory inhaled corticosteroids to address the inflammatory process in the airways (maintenance) and bronchodilators (relievers) for relief of the bronchospasm. Many studies have shown that asthma mortality is linked to poor use of anti-inflammatory inhaler treatment and over-reliance on short- acting β2 bronchodilator reliever therapy to treat asthma exacerbations. In many LMICs including South Africa, the use of controller treatment use of anti-inflammatory inhalers is limited, with only 40% of people with severe asthma symptoms using regular ICS for chronic asthma treatment, but with over 89% using their short-acting β2 agonists. There is a large body of evidence showing that overuse of SABAs is linked with asthma mortality and poorer outcomes.

The combination treatment with budesonide/formoterol for the management of asthma has transformed asthma treatment in high-income countries (HIC), where it is recommended in the very first step of asthma treatment as both an anti-inflammatory and reliever therapy. With the "as needed" use of budesonide/formoterol, asthmatics benefit from the additional dose of a maintenance anti-inflammatory dose, which improves symptom control and reduces exacerbations. This approach has not been adopted in many LMICs related to access to budesonide/formoterol and its cost and therefore, people in LMICs are relegated to use of Track 2 of Global Initiative of Asthma (GINA) treatment which still suggests the use of separate anti-inflammatory and reliever inhalers.

To address this gap, a large body of randomized controlled clinical trial evidence (SYGMA, Novel START, PRACTICAL, and several trials of SMART), have shown that use of budesonide/formoterol as needed (for exacerbations) and for long-term controller treatment compared to separate inhaled corticosteroid and short-acting bronchodilators, reduces the number of asthma exacerbations and improves quality of life. The trials have though been limited in that there is no data on the cost-effectiveness of this approach in lower resourced settings and limited data from small studies participant numbers (<100) of this approach in children 6-11 years of age. Based on this, the approach of using budesonide/formoterol has not been recommended by the Global Initiative of Asthma (GINA) strategy for global asthma management in Step 1 and 2 of treatment in children 6-11 years of age both in HIC and LMICs, but rather on the higher steps of asthma treatment where symptoms are more severe.

The investigators therefore propose in a randomized controlled trial to assess the efficacy of budesonide/formoterol compared to the standard of care (separate inhaled corticosteroid and bronchodilator) inhaler approach to prevent asthma exacerbations, improve asthma control and quality of life and to also assess the cost-effectiveness of budesonide/formoterol compared to standard of care in children and adolescents in South Africa. The data will be novel as the investigators will for the first time include a large number of children in a clinical trial comparing the two approaches, to provide definitive evidence of the efficacy and cost-effectiveness of this approach in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age for inclusion children and adolescents 6-18 years at the time of consent
* Known asthmatic on treatment.
* Newly diagnosed asthma based on investigator review and/or medical report.
* All patients will have their asthma diagnosis confirmed (both new or known asthmatic patients) by either spirometry with reversibility or excessive diurnal variability by PEFR twice daily over 2 weeks.
* Ability to perform Peak Expiratory Flow rate and/or bronchodilator reversibility testing.
* Only participants with mild, or moderate asthma , based on medical history
* At least one exacerbation of asthma in the past year as defined by an event requiring treatment with systemic corticosteroids for ≥3 days and/or a hospitalisation/emergency room visit for asthma requiring treatment with systemic corticosteroids.
* Written consent from the participant or parent/guardian and assent from study participants where applicable.
* Participant and/or parent/guardian agrees to comply with the study procedures, including the completion of the visits and be available for contact for telephonically for the non-contact visits

Exclusion Criteria:

* Tuberculosis (TB): active TB disease and contact with people with active TB disease in the last 6 months.
* Chronic sputum expectoration, chest pain, shortness of breath, dizziness, or light-headedness in the last 2 months.
* Cardiac arrythmia.
* Chronic conditions: thyrotoxicosis, phaeochromocytoma, cardiovascular disease, severe hypertension.
* Uncontrolled diabetes mellitus
* Patients with Peak Expiratory Flow Rate < 50% of predicted , as these would be classified as severe asthmatics.
* Patients with any history of life-threatening asthma, defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s).
* Any use of biological therapy or immunomodulatory therapy such as methotrexate or regular oral prednisolone for the asthma management (STEP 5 GINA therapy).
* Any surgical or medical condition that would significantly alter the absorption, distribution, metabolism or excretion of the IMP which may jeopardise the safety of the participants. The investigator should make this determination in consideration of the volunteer's medical history.
* Any physical, mental or social condition, laboratory abnormality of history of illness that in the investigator's judgement might jeopardise the safety of the participant in the context of the study or might interfere with study procedures or the ability of the participant to adhere to and complete the study. The investigator should make this determination consideration of the volunteer's medical history.
* Inability to present for follow-up or leaving the study area within 12 months of enrolment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1038 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbations in 52 weeks ( End of study) | 52 weeks
  Questionnaire- based-tool to capture number of exacerbations will be administered biweekly via a short message system, 6 monthly telephonic consultations and alternative 6 monthly clinic visits. Unscheduled visits will be captured using the bi-weekly questionnaires.

SECONDARY OUTCOMES:
Cost effectiveness | 52 weeks
  Cost effectiveness will assessed using health economics , health facility and quality of life questionnaires that will be administered to the participants, caregivers and facility managers.

CONTACTS AND LOCATIONS:
Overall Officials: Limakatso Lebina, PhD, Study Director — Africa Health Research Institute
Locations (1):
- Africa Research Health Institute Clinical Trial Unit, Mtubatuba, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
A dissemination plan will be developed with all project partners prior to study completion. After study completion, results will be disseminated using the following strategies: written methods (i.e., publications in peer reviewed scientific journals), presentations at scientific conferences and workshops, in person dissemination of results to the research participants, the ministry of health and using electronic methods such as the project website and electronic media to publish results.
Supporting Information: Study Protocol
Time Frame: 3 years for the time of request
Access Criteria: A log of names, signatures and initials of all staff authorised to enter data into a participant's clinic file and eCRF will be kept.

REFERENCES:
- [Derived] Hlophe ST, Ndimande NN, Ngobese N, Mkwanazi E, Bird K, Mbonigaba J, Otwombe K, Lebina L, Mortimer K, Masekela R. Anti-inflammatory reliever therapy for asthma using inhaled budesonide/formoterol as-needed with or without maintenance in South African children (AIR-SA 001): a description of a randomised clinical trial protocol. BMJ Open Respir Res. 2025 Nov 17;12(1):e003378. doi: 10.1136/bmjresp-2025-003378. PMID 41253413

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT06429475/Prot_SAP_ICF_000.pdf